CLINICAL TRIAL: NCT07064590
Title: Investigation of Frontopolar Transcranial Magnetic Stimulation on Correlates of Craving in Alcohol Addiction
Brief Title: Effects of Frontopolar TMS in Alcohol Craving
Acronym: TMS-SUD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Jonathan Repple, Prof. Dr., Goethe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-2021
Record Dates: First submitted 2025-06-06; First posted 2025-07-14 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Addiction
Keywords: frontopolar transcranial magnetic stimulation (TMS); craving; alcohol addiction; addiction treatment; virtual reality (VR); magnetic resonance imaging (MRI); Continuous Theta Burst Stimulation (cTBS); neuromodulation; structural and functional brain connectivity; connectome; neurophysiological craving markers; prediction; physiological craving markers; psychological craving markers; Neuronavigation
MeSH Terms: conditions — Alcoholism | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Frontopolar cTBS Intervention (Experimental): Participants in this arm will receive 15 sessions of continuous theta burst stimulation (cTBS) over the left frontopolar cortex across 5 consecutive days (3 sessions/day) using neuronavigation based on individual MRI. The stimulation intensity is set at 110% of the resting motor threshold. Virtual Reality Cue Exposure and Craving Assessment (VR-CECA) and psychological craving assessment will be performed before and after the TMS intervention. Baseline structural and functional MRI scans will be acquired before stimulation for brain connectivity analysis.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Patients will receive cTBS, a five-minute protocol with inhibitory effects over the left frontal pole, using an accelerated design comprising three sessions daily for five consecutive days (15 sessions total). Stimulation will be delivered using a Magventure TMS device routinely used in clinical practice at the Department of Psychiatry, Psychotherapy and Psychosomatics, University Hospital Frankfurt. TMS is generally well tolerated, with mild headache or scalp discomfort as common side effects. Localization will be based on individual MRI data: after cortical parcellation with FreeSurfer 7.4.1, the left frontal pole centroid will be extracted. Coil placement will be neuronavigated using the Localite Neuronavigator. Stimulation will be applied at 110% resting motor threshold (rMT; 3-pulse bursts at 50 Hz, 5 Hz interburst; 1800 pulses/train; 60 s intertrain). Intensity may be gradually increased until 110% rMT is reached.

SUMMARY:
The goal of this interventional study is to learn if continuous theta burst stimulation (cTBS) applied over the left frontopolar cortex can reduce psychological, physiological, and neurobiological markers of alcohol craving in patients with alcohol dependence (AD).

The main questions it aims to answer are:

* Does cTBS over the left frontopolar cortex reduce psychological and physiological measures of alcohol craving in individuals with AD?
* Are baseline structural and functional brain connectivity patterns associated with individual differences in cTBS-induced changes in craving?

The participants will:

* Receive cTBS over the left frontopolar cortex using an accelerated protocol comprising 15 TMS-sessions on five consecutive days
* Undergo psychological and physiological assessments of alcohol craving before and after the TMS intervention
* Complete magnetic resonance imaging (MRI) sessions to assess baseline brain structural and functional connectivity

This study aims to advance the understanding of the neurophysiological mechanisms underlying craving in AD and the identification of potential biomarkers for predicting psychological and physiological craving reductions.

DETAILED DESCRIPTION:
Alcohol dependence (AD) is a prevalent and debilitating condition characterized by a chronic inability to control alcohol consumption despite adverse consequences. Current treatment options have limited efficacy, highlighting the pressing need for innovative approaches. Continuous Theta Burst Stimulation (cTBS) is a form of transcranial magnetic stimulation (TMS) that has shown promise in modulating brain activity associated with craving and addiction.

This study aims to explore the effects of cTBS applied over the left frontopolar cortex on psychological, physiological, and neurobiological markers of alcohol craving in patients with AD. Specifically, this study will assess TMS-induced changes in psychological alcohol craving using the Penn Alcohol Craving Scale (PACS), and physiological alcohol craving using physiological craving markers, including heart rate (HR), skin temperature (ST) and skin conductance (SC), and their changes during Virtual Reality Cue Exposure and Craving Assessment (VR-CECA) before and after the TMS intervention. Additionally, the study aims to explore the relationship between neurobiological craving markers utilizing baseline structural and functional brain connectivity as assessed by magnetic resonance imaging (MRI) and TMS-induced changes in psychological and physiological alcohol craving.

This study aims to include a total of 34 patients aged 18-65 years with an ICD-10 diagnosis of AD. All participants undergo 15 sessions of accelerated cTBS targeting the left frontopolar cortex over five consecutive days using neuronavigation based on individual MRI scans. Clinical (questionnaires, diagnostic interviews) and behavioural (VR-CECA) assessments are conducted at two time points: pre-TMS intervention and post-TMS intervention. Structural and functional MRI scans are acquired before the TMS intervention to assess individual brain connectivity.

The primary outcome will be the TMS-induced change in psychological alcohol craving assessed with the PACS. Secondary outcomes include TMS-induced changes in physiological craving markers (HR, ST, and SC) during VR-CECA and TMS-induced changes and psychopathological states that will be assessed through a battery of clinical questionnaires.

This study hypothesizes that frontopolar cTBS will reduce psychological and physiological alcohol craving in patients with AD. Additionally, this study expects that baseline structural and functional connectivity will predict TMS-induced changes in physiological alcohol craving, providing insights into individual brain network variability on the effect of frontopolar cTBS.

This study aims to advance the understanding of the neurophysiological mechanisms underlying craving in AD and the identification of potential biomarkers for predicting psychological and physiological craving reductions. If successful, this could lead to more targeted and effective interventions for AD, ultimately improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18-65
* ICD-10 diagnosis of alcohol dependence
* Ability to give consent
* Sinus rhythm in ECG

Exclusion Criteria:

* Current psychotic symptoms in patients with psychotic disorders (F20, F23, F10.5)
* Contraindication against TMS or MRI
* Severe neurological disorders such as epilepsy, stroke, neuroinflammatory disorders (e.g., multiple sclerosis). A history of seizures only in the context of alcohol withdrawal does not represent a contraindication, unless the seizure happened in the last 3 weeks before study inclusion.
* Acute withdrawal symptoms (CIWA-Ar > 5)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
TMS-induced changes in psychological alcohol craving assessed with the Penn Alcohol Craving Scale (PACS) | The PACS will be assessed at baseline before the start of the TMS Intervention (Pre-TMS, Day 0) and after the final TMS session (post-TMS, Day 5)
  The primary outcome measure is the TMS-induced changes in psychological craving intensity. Self-reported psychological alcohol craving as measured by the Penn Alcohol Craving Scale (PACS) will be assessed before the frontopolar TMS intervention (pre-TMS at baseline) and after the final frontopolar TMS session (post-TMS). The PACS is a five-item, self-report measure that includes questions about the frequency, intensity, and duration of craving, the ability to resist drinking, and asks for an overall rating of craving for alcohol for the previous week. Each question is scored on a scale of 0 to 6. The mean total score across the five items (range 0-6) will be calculated, with higher scores indicating greater craving. In exploratory analyses, individual PACS items can also be examined separately to capture distinct dimensions of craving (e.g., frequency, intensity, or duration).

SECONDARY OUTCOMES:
TMS-induced change in heart rate (BPM) during virtual reality alcohol cue exposure | HR is continuously recorded during VR alcohol cue exposure sessions conducted on Day 1 (prior to the first TMS session) and Day 5 (following the final TMS session), allowing assessment of TMS-induced changes in physiological craving response.
  TMS-related changes in heart rate (HR; beats per minute) during VR-based alcohol craving induction will be assessed. HR is continuously recorded throughout each VR cue exposure session. For each session, the difference in minimum and maximum HR (within-session change) will be calculated as an index of physiological craving reactivity. These within-session changes are then compared between sessions (Day 1 → Day 5) to evaluate TMS-induced modulation of HR responses. Further indices that can be derived from this assessment are mean, maximum, and minimum HR.
TMS-induced change in skin conductance (µS) during Virtual reality alcohol cue exposure | SC is continuously recorded during VR alcohol cue exposure sessions conducted on Day 1 (prior to the first TMS session) and Day 5 (following the final TMS session), allowing assessment of TMS-induced changes in physiological craving response.
  TMS-related changes in skin conductance (SC; µS) will be assessed during VR-based alcohol craving induction. SC is continuously recorded throughout each VR cue exposure session. For each session, the difference in minimum and maximum SC (within-session change) will be calculated as an index of physiological craving reactivity. These within-session changes are then compared between sessions (Day 1 → Day 5) to evaluate TMS-induced modulation of SC responses. Further indices that can be derived from this assessment are mean, maximum, and minimum SC.
TMS-induced change in skin temperature (°C) during Virtual reality alcohol cue exposure | ST is continuously recorded during VR alcohol cue exposure sessions conducted on Day 1 (prior to the first TMS session) and Day 5 (following the final TMS session), allowing assessment of TMS-induced changes in physiological craving response.
  TMS-related changes in skin temperature (ST; °C) are assessed during VR-based alcohol craving induction. ST is continuously recorded throughout each VR cue exposure session. For each session, the difference in minimum and maximum ST (within-session change) will be calculated as an index of physiological craving reactivity. These within-session changes are then compared between sessions (Day 1 → Day 5) to evaluate TMS-induced modulation of ST responses. Further indices that can be derived from this assessment are mean, maximum, and minimum ST.
TMS-induced change in self-reported craving during VR exposure using Visual Analogue Scale (VAS) | Day 1 (pre-TMS; pre-VR and post-VR) and Day 5 (post-TMS; pre-VR and post-VR)
  TMS-related changes in subjective craving ratings will be measured before and after each VR alcohol cue exposure. Participant reactivity during VR alcohol cue exposure is assessed using a 10-item Visual Analog Scale (VAS; 0-100). Items measure both general affective/physiological states (e.g., tension, stress, feeling challenged, control) and alcohol-related urges (e.g., thoughts, desire, craving for alcohol). Each item is rated from 0 ("not at all") to 100 ("very"/"strong"). The mean score across all 10 items will be calculated. Additionally, individual item scores will be calculated separately to investigate item-specific/domain-specific changes. VAS ratings are obtained immediately before and immediately after each VR session to assess changes in reactivity following alcohol cue exposure. Additionally, VAS rating assessed before the TMS intervention and after the final TMS session will be compared to assess TMS-related changes in craving reactivity.
TMS-induced change in self-reported craving assessed with the Mannheimer Craving Scale (MaCS) | The MaCS will be assessed at baseline before the start of the TMS Intervention (Pre-TMS, Day 0) and after the final TMS session (post-TMS, Day 5)
  Changes in self-reported psychological alcohol craving will be assessed using the Mannheimer Craving Scale (MaCS) before and after the frontopolar TMS intervention. The MaCS measures obsessive-compulsive symptoms related to substance use and dependence. It includes 12 core items and 4 additional items. Each of the 12 core items is rated on a 5-point Likert scale (0-4), with higher values indicating greater symptom intensity. The four additional items include three visual analog scales (VAS; 0-100) assessing average craving intensity, maximum craving intensity, and craving frequency during the past seven days, as well as one item assessing duration of abstinence (in days). The mean total score of the 12 core items (range: 0-4) will be computed. VAS measures and abstinence duration will be analyzed separately as supplementary indicators of craving. Exploratory analysis could also include the calculation of mean scores of subscales.
TMS-induced change in self-reported psychological craving assessed by the Craving-Automatized-Scale-Alcohol (CAS-A) | The CAS-A will be assessed at baseline before the start of the TMS Intervention (Pre-TMS, Day 0) and after the final TMS session (post-TMS, Day 5)
  The CAS-A is a 15-item self-report questionnaire that assesses situations of loss of control or automatic drinking, and is here implemented to evaluate changes in self-reported psychological craving before and after TMS intervention. Each item is rated on a 6-point Likert scale (0 = "never" to 5 = "always"), referring to the participant's most recent drinking episode within the last 7 days. Item 16 records when the participant last consumed alcohol. The mean total score across all 15 items will be calculated. Additionally, further mean subscale scores (e.g., 5 CAS-A factors as "only aware in hindsight," "no deliberate decision," "contrary to intention," "no perception," and "no control"; or 2 factors, "unaware" and "nonvolitional.") will be used to explore distinct dimensions of craving and drinking behavior.
Correlation between baseline brain connectivity and changes in heart rate (BPM) increase during VR | MRI and, therefore, structural and functional connectivity is assessed at baseline (Day 0) and heart rate change during VR sessions before TMS intervention (Day 1) and after the final TMS intervention (Day 5)
  Correlation between baseline structural or functional brain connectivity (as assessed via MRI prior to TMS) and the increase in heart rate during VR craving induction. Connectivity data are derived using diffusion-weighted imaging and resting-state fMRI, processed via CATO and analyzed using network-based statistics.
TMS-induced changes in clinician-reported depressive symptoms using the MADRS | The MADRS will be assessed at baseline before the start of the TMS Intervention (Pre-TMS, Day 0) and after the final TMS session (post-TMS, Day 5)
  Changes in self-reported craving levels will be measured before and after the 5-day TMS intervention, assessed with the Montgomery-Åsberg Depression Rating Scale (MADRS), is a 10-item, clinician-administered scale to assess depression severity. It rates symptoms like sadness, feelings of emptiness, tension, and reduced interest, with scores from 0 to 6 for each item, resulting in a total score from 0 to 60. Higher scores indicate more severe depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Repple, Prof. Dr., Principal Investigator — Klinik und Poliklinik für Psychiatrie, Psychosomatik und Psychotherapie Universitätsklinikum Frankfurt; Mathias Luderer, Dr. med., Principal Investigator — Klinik und Poliklinik für Psychiatrie, Psychosomatik und Psychotherapie Universitätsklinikum Frankfurt; Maren Schmidt-Kassow, Prof. Dr., Principal Investigator — Klinik und Poliklinik für Psychiatrie, Psychosomatik und Psychotherapie Universitätsklinikum Frankfurt
Locations (1):
- Klinik und Poliklinik für Psychiatrie, Psychosomatik und Psychotherapie Universitätsklinikum Frankfurt, Goethe-Universität, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Williams JB, Kobak KA. Development and reliability of a structured interview guide for the Montgomery Asberg Depression Rating Scale (SIGMA). Br J Psychiatry. 2008 Jan;192(1):52-8. doi: 10.1192/bjp.bp.106.032532. PMID 18174510
- [Background] Nakovics H, Diehl A, Geiselhart H, Mann K. [Development and validation of an overall instrument to measure craving across multiple substances: the Mannheimer Craving Scale (MaCS)]. Psychiatr Prax. 2009 Mar;36(2):72-8. doi: 10.1055/s-2008-1067546. Epub 2008 Oct 15. German. PMID 18924060
- [Background] Flannery BA, Volpicelli JR, Pettinati HM. Psychometric properties of the Penn Alcohol Craving Scale. Alcohol Clin Exp Res. 1999 Aug;23(8):1289-95. PMID 10470970
- [Background] Vollstadt-Klein S, Lemenager T, Jorde A, Kiefer F, Nakovics H. Development and validation of the craving automated scale for alcohol. Alcohol Clin Exp Res. 2015 Feb;39(2):333-42. doi: 10.1111/acer.12636. PMID 25684052